CLINICAL TRIAL: NCT02916680
Title: Pancreatic Islet Transplantation in the Anterior Chamber of the Human Eye - a Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Eye ITPL
Record Dates: First submitted 2016-03-31; First posted 2016-09-27 (Estimated); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Pancreatic islet transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Islets of Langerhans Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pancreatic islet transplantation (Experimental): Pancreatic islet transplantation in the anterior chamber of the human eye
  Interventions: Procedure: Pancreatic islet transplantation in the anterior chamber

INTERVENTIONS:
Procedure: Pancreatic islet transplantation in the anterior chamber — Transplantation of allogeneic pancreatic islet cells into the anterior chamber of a severely visual impaired diabetic human eye

SUMMARY:
The overall objective is to establish that transplantation of allogeneic pancreatic islet cells into the anterior chamber of a severely visual impaired diabetic human eye is safe and does not cause ophthalmic or systemic complications. Furthermore, the change in insulin production, glucose control and hypoglycaemia awareness will be assessed.

DETAILED DESCRIPTION:
Investigators intend to transplant 4 Type 1 Diabetes mellitus patients with compromised vision in one or both eyes due to diabetic or other complications, and who have already received kidney transplantation (i.e., already on immunosuppression). Transplantation of allogeneic pancreatic human islets will be performed into the anterior chamber of a single eye with compromised vision. Since the recipients are already immunosuppressed due to maintenance therapy for the kidney graft, investigators will only use non-steroidal anti-inflammatory drug (NSAID).

Only in case of uncontrolled reaction, steroid should be used under guidance of the ophthalmologists. Investigators will neither inject local immunosuppressive drugs nor change ongoing immunosuppressive medication in the pilot study.

The overall objective is to establish that transplantation of allogeneic pancreatic islet cells into the anterior chamber of a severely visual impaired diabetic human eye is safe and does not cause ophthalmic or systemic complications. Furthermore, the change in insulin production, glucose control and hypoglycaemia awareness will be assessed.

In this pilot study investigators aim to gain experience in the technique, to obtain preliminary data on the amount of insulin that can be expected per transplanted islet equivalent (IEQ) and observe possible local reactions. These data will help to design a future larger study in patients without visual impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 Diabetes (American Diabetes Association criteria)
2. Kidney transplant recipient with ongoing immunosuppression
3. At least one eye with extensive loss of vision from hand motion to no light perception due to damage of retina or optic nerve
4. Age ≥ 18 years
5. Normal cornea with good visualization of the anterior segment
6. Patient not eligible or with no wish for standard pancreatic islet into the hepatic portal system or pancreas transplantation

Exclusion Criteria:

1. Uncontrolled diabetic retinopathy
2. Signs of current infection
3. Poor visualization of the anterior chamber

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2016-03; Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Absence of ophthalmic complications | 90 days
  safety

SECONDARY OUTCOMES:
Change in insulin production | 90 days
  Change in insulin production as derived from change in C-peptide, insulin, pro-insulin and glucose levels during the mixed meal tolerance test (MMTT) at Day 90 compared to baseline
Change in insulin requirements | 90 days
  Change in insulin requirements: 3-day average daily insulin dose at baseline compared to Day 90 (Day 87 through Day 89)
Change in HbA1c | 90 days
  Change in HbA1c levels from baseline (Day 0 pre-transplant) at Day 90
Change in fasting glucose | 90 days
  Change in fasting glucose from baseline (Day 0 pre-transplant) at Day 90
Change in total number of hypoglycemic events | 90 days
  Change in total number of hypoglycemic events 3-day average at baseline compared to Day 90 (Day 87 through Day 89) as assessed by continuous glucose monitoring (CGMS)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Y Donath, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No